CLINICAL TRIAL: NCT04208984
Title: Interactive Multimedia Diversion Device With Breath Control
Brief Title: Diversion Device With Breath Control
Status: Not yet recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Ben Chortkoff, Professor, University of Utah
Other Study IDs: 104924
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Induction of Anesthesia
Keywords: induction; anesthesia; children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Patients randomized to this group will receive standard of care induction of anesthesia
- Study: Patients randomized to this group will receive induction of anesthesia using the Lullabreath game
  Interventions: Device: Study
- Music Video: Patients randomized to this group will receive induction of anesthesia using the music video game
  Interventions: Other: Music Video

INTERVENTIONS:
Device: Study — After consent and assent the child and parent will be introduced the Lullabreath in pre-op. The purpose of Lullabreath will be explained and the Lullabreath will be taught (15 minutes). The parent will complete the PROMIS Proxy Anxiety short form. The children are then taken to the operating room (leave parents) with the Lullabreath. The anesthesiologist will hook the device up to the anesthesia circuit and start the Lullabreath. The child will then undergo induction of anesthesia while playing the Lullabreath.
  Groups: Study
Other: Music Video — After consent and assent the child and parent will be introduced to the game in pre-op. The purpose of the game will be explained and the game will be taught (15 minutes). The parent will complete the PROMIS Proxy Anxiety short form. The children are then taken to the operating room (leave parents) with the game. The anesthesiologist will hook the device up to the anesthesia circuit and start the game. The child will then undergo induction of anesthesia while playing the game. The child can choose to watch one of two music videos (Frozen, Lion King)
  Groups: Music Video

SUMMARY:
The experience for many children who need to undergo anesthesia induction by breathing anesthetic vapors in the operating room is frightening to the child. We have developed a computer-based game system that uses breathing-in and breathing-out as a game controller. We believe that the immersive game experience will encourage breathing patterns ideal for anesthetic induction while providing fun and diversion for the child, lessening or eliminating the fear that typically accompanies breathing anesthetics.

The purpose of the study is to determine whether diversion and breathing encouragement offered by a game and this device

DETAILED DESCRIPTION:
Anesthetic induction in children often requires pre-induction administration of pharmacologic sedatives to directly soothe the anxiety of the child (patient) as well as indirectly soothe the vicarious anxiety of the parents. The sterile, foreign environment, the parade of unfamiliar uniformed health-care workers, the sober weightiness of the adults' in their approach to the preparation for surgery, and the often cold, loud, and different smelling environment all contribute to an escalating level of anxiety. This anxiety manifests as a fear of separation (between child and parent) and a physiologic elevation in catecholamine release (fight or flight response: tachycardia, tachypnea, hypertension, sweating, crying, and escape behavior).

Pharmacologic sedatives are effective but have substantial drawbacks. They may be challenging to administer. They are distasteful and/or uncomfortable for the children to receive. They frequently have half-lives that extend beyond the length of surgery. They require 30 minutes to one-hour to take full effect. And, they may lead to more confusion or delirium upon emergence.

Distraction by the anesthesiologist, whether through storytelling, by entertaining with humor, by singing to the child, or by utilizing a computer, phone, or tablet device to provide games or videos, has been an effective tool and/or alternative to pharmacologic sedation for children to help smooth the experience of separation and the experience of undergoing anesthetic induction.1-3 In contrast to children, induction of anesthesia in adults is routinely accomplished by administration of intravenous medications. The intravenous route provides the most rapid and least sensory repugnant initiation of anesthesia. Starting an intravenous line in an awake child can be technically challenging for the physician and emotionally frightening and physically painful for the child. Because of that, for elective pediatric surgeries, the anesthesiologist often opts to initiate anesthesia in children by having the child breath anesthetic vapors (inhalation induction). Inhalation induction is dependent on the breathing of the patient for medication delivery. When children are anxious they often "breath-hold" and fight to avoid the anesthetic delivery circuit when presented with an anesthetic mask. This not only delays and complicates anesthetic delivery, it is uncomfortable and frustrating experience for the patient and for the anesthesiologist, and emotionally uncomfortable for the operating room health care team to observe. Providing a child with a non-frightening motivation to breathe through the facemask and anesthesia circuit would speed the delivery of anesthetic during induction and improve the experience for all involved. In addition, induction of anesthesia in adults is almost always preceded with a two to four minute "pre-oxygenation" period during which time the adult breathes 100% oxygen through the facemask and anesthetic circuit. The intent is to exchange the residual air in the lungs (the functional reserve capacity) with oxygen, providing a physical reservoir of life-extending oxygen should ventilating or intubating the patient prove difficult. This safety measure is not practical in children since they often reject breathing through the mask. If breathing through the mask was seen as an enjoyable aspect of a game rather than as a frightening preliminary step toward surgery, children might participate in pre-oxygenation thereby increasing the safety margin during induction of anesthesia.

We are creating an inexpensive gaming system that would provide an immersive distraction and would simultaneously encourage effective breathing through the anesthesia circuit by combining selected or original computer games with an engineered adaptor that turns breathing into the game controller.

A respiratory flow sensor is connected to a laptop computer and controls a simple computer game, where, e.g., a rocket ship flying through space can be made to swerve to the left or the right, depending on how much the subject inhales or exhales. The goal of the game is to collect virtual 'coins' by steering the rocket ship through them. The computer game is designed to keep the subject engaged and motivates the subject to breathe through the mask. During an initial phase at the very beginning of the game, the software detects the normal level of the subject's breathing. During the actual game the 'coins' are spaced in the game to ensure that the subject's breathing does not deviate by more than +-30% from their normal breathing level.

Except for the flow-sensor, which is connected in-line between the standard face mask and the standard breathing circuit, the anesthetic equipment is the same that is routinely used on patients. The system does not display any respiratory measurements to the anesthesia provider taking care of the patient and no clinical or dosing decisions are based on the system's involvement or output. The system does record the breathing signals in an internal file for later off-line analysis, but that data is de-identified and not made available to the clinician taking care of the subject.

ELIGIBILITY:
Inclusion Criteria:

* 4-11 year old children undergoing anesthesia for any procedure

Exclusion Criteria:

* Visual impairment
* non english speaking
* Premature infants
* children previously exposed to the chemotherapeutic agent bleomycin

Ages: 4 Years to 11 Years | Sex: All
Age Groups: Child
Study Population: 4-11 year old children undergoing anesthesia for any procedure without visual impairment, non english speaking, Premature infants and children previously exposed to the chemotherapeutic agent bleomycin
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Administered to parents directly after induction of anesthesia
  Anxiety measured by the PROMIS Anxiety Parent-Proxy questionnaire, minimum 0, maximum 100 points (t-score), higher score means higher anxiety
End-tidal oxygen at the beginning of anesthesia | Measured directly after induction
  End-tidal oxygen concentration measured at the start of anesthesia
Anxiety | Administered to the anesthesiologist caring for the patient directly after induction of anesthesia
  Anxiety measured by the PROMIS Anxiety Parent-Proxy questionnaire, minimum 0, maximum 100 points (t-score), higher score means higher anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Kai Kuck, PhD, Study Chair — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No